CLINICAL TRIAL: NCT03133559
Title: Mapping the Human Immunodeficiency Virus Chronobiome, (HIV)
Brief Title: Mapping the Human HIV Chronobiome
Acronym: HCB
Status: Suspended | Type: Observational
Why Stopped: Protocol Modification is pending
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Carsten Skarke, MD, Research Assistant Professor, University of Pennsylvania
Other Study IDs: 825626
Record Dates: First submitted 2016-12-21; First posted 2017-04-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hiv; Healthy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen = None for Cohort 1. Completed Cohort 1.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1: Patients infected with HIV off antiretroviral therapy
  Interventions: Other: Observational
- Cohort 2: Patients infected with HIV experiencing virologic control, but with blunted immunologic recovery
  Interventions: Other: Observational
- Cohort 3: Matched healthy volunteers
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — We will use a deep phenotyping approach to collect multidimensional datasets from individuals infected with HIV compared to healthy controls to define circadian rhythm disruptions associated with HIV infection.

SUMMARY:
Individuals infected with HIV have a high risk of developing metabolic comorbidities not traditionally associated with the immune dysregulation and deficiency associated with HIV infection and AIDS. Many of these comorbidities in HIV uninfected individuals have been linked to a disordered circadian clock function. The study investigators will further evaluate the circadian clock in HIV infection as a mechanism underlying the metabolic dysregulation in this population.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Diagnosis of HIV infection with CD4+ counts <500 cells/mm3 while untreated;
* Cohort 2: Diagnosis of HIV infection with CD4+ counts <300 cells/mm3 on ARV;
* Cohort 3: Volunteers must be in good health as based on medical history, physical examination, vital signs, and laboratory tests as deemed by PI;
* Volunteers are capable of giving informed consent;
* 25-50 years of age;
* Own a smartphone which installs the remote sensing applications;
* Non-smoking;
* Male subjects only if feasible during recruitment; and
* In case female volunteers are invited to enroll: non-pregnant, female subjects must consent to a urine pregnancy test.
* Females of child bearing potential will be asked to use a medically accepted method of birth control (such as oral contraceptives, intra-uterine device (IUD), or condom with spermicide) while you participate in the study.
* The use of contraception will NOT be required for male participants.

Exclusion Criteria:

* Recent travel across more than two (2) time zones (within the past month);
* Planned travel across more than two (2) time zones during the planned study activities;
* Volunteers with irregular work hours, e.g. night shifts or becoming a parent;
* Use of illicit drugs;
* High dose vitamins (Vitamin A, Vitamin C, Vitamin E, Beta Carotene, Folic Acid and Selenium), alcohol and any over-the counter NSAID in the (2) two weeks before the start of the 48 hour deep phenotyping period (Females who are taking birth control pills can continue so for the duration of this study).;
* History of abdominal surgery;
* Subjects, who have received an experimental drug, used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening;
* Subjects with any abnormal laboratory value or physical finding that according to the investigator may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject.
* Women who are breastfeeding.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cohort 1: patients infected with HIV off antiretroviral therapy;
  Cohort 2: patients infected with HIV experiencing virologic control, but with blunted immunologic recovery;
  Cohort 3: matched healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Time-of-day fluctuations in core clock gene expression | 48 hours
  Relative expression normalized to housekeeping genes (GAPDH, ACTB) plotted by time of day (morning, afternoon, evening, night with target times of 08:00, 14:00, 20:00, 02:00 +/- 1 hour)

SECONDARY OUTCOMES:
Variance explained [R^2 values] | 48 hours
  To evaluate the linear relationships between every pairwise combination of variables in the integrated dataset, the R^2, or coefficient of determination, will be calculated for each pair using linear regression. A heat map of the proportion of variance in each variable (e.g. mobility, light exposure, systolic blood pressure) explained by each other variable will then be constructed to allow an integrative exploration of these data. This approach allows to integrate multiple measurements with different units of measure. The measurements include communication (number of phone calls and text messages), mobility (miles traveled), light exposure, blood pressure, heart rate, heart rate variability, sleep/wake times, body core temperature, multiomics outputs (abundance of metabolites, proteins, microbiota) and markers of cellular and inflammatory function and disease state (HIV infection).
Variance explained [R^2 values] | up to 4 months
  To evaluate the linear relationships between every pairwise combination of variables in the integrated dataset, the R^2, or coefficient of determination, will be calculated for each pair using linear regression. A heat map of the proportion of variance in each variable (e.g. mobility, light exposure, systolic blood pressure) explained by each other variable will then be constructed to allow an integrative exploration of these data. This approach allows to integrate multiple measurements with different units of measure. The measurements include communication (number of phone calls and text messages), mobility (miles traveled), light exposure, and sleep/wake times.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Skarke, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Institute for Translational Medicine and Therapeutics (ITMAT), University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
To be determined